CLINICAL TRIAL: NCT05446740
Title: A Phase 1 Randomized, Observer-blind, Dose-escalation Study to Evaluate the Safety, Reactogenicity and Immunogenicity of an mRNA-based Monovalent Influenza Vaccine Candidate in Healthy Younger and Older Adults
Brief Title: A Study on the Safety, Reactogenicity and Immune Response of a Vaccine Against Influenza in Healthy Younger and Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 217895; 2022-000489-17 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Influenza, Human
Keywords: Influenza; Safety; Reactogenicity; Immunogenicity; mRNA vaccine; Healthy younger adults; Healthy older adults
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be observer-blind with regards to the study intervention and open-label with regards to the dose level for participants and investigators and open-label for the sponsor. For dose cohorts 6, 7, 10 and 11 the study will be single-blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- YA GSK4382276A Dose level 1 Group (Experimental): Eligible young adults (YA) participants receive dose level 1 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 1
- YA GSK4382276A Dose level 2 Group (Experimental): Eligible young adults (YA) participants receive dose level 2 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 2
- YA GSK4382276A Dose level 3 Group (Experimental): Eligible young adults (YA) participants receive dose level 3 GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 3
- YA GSK4382276A Dose level 4 Group (Experimental): Eligible young adults (YA) participants receive dose level 4 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 4
- YA GSK4382276A Dose level 6 Group (Experimental): Eligible YA participants receive dose level 6 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 6
- YA GSK4382276A Dose level 7 Group (Experimental): Eligible YA participants receive dose level 7 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 7
- YA GSK4382276A Dose level 8 Group (Experimental): Eligible YA participants receive dose level 8 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 8
- YA GSK4382276A Dose level 9 Group (Experimental): Eligible YA participants receive dose level 9 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 9
- YA GSK4382276A Dose level 10 Group (Experimental): Eligible YA participants receive dose level 10 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 10
- YA GSK4382276A Dose level 11 Group (Experimental): Eligible YA participants receive dose level 11 of GSK4382276A study intervention administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 11
- YA Control 1 Group (Active Comparator): Eligible YA participants receive single dose of FDQ21A-NH administered at Day 1.
  Interventions: Combination Product: FDQ21A-NH
- YA Control 2 Group (Active Comparator): Eligible YA participants receive single dose of FDQ22A-NH administered at Day 1.
  Interventions: Combination Product: FDQ22A-NH
- OA GSK4382276A Group (Experimental): Eligible OA participants receive single dose of GSK4382276A study intervention at 1 dose level selected from the first 3 dose levels in YAs, administered at Day 1.
  Interventions: Biological: GSK4382276A Dose level 1; Biological: GSK4382276A Dose level 2; Biological: GSK4382276A Dose level 3
- OA Control Group (Active Comparator): Eligible OA participants receive single dose of FDQ21A-NH administered at Day 1.
  Interventions: Combination Product: FDQ21A-NH

INTERVENTIONS:
Biological: GSK4382276A Dose level 1 — Dose level 1 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A Dose level 1 and OA GSK4382276A Selected Dose level from YA groups, at Day 1. Potential intermediate dose levels may be evaluated, with the total number of dose levels per age group not exceeding 5.
  Other Names: Flu mRNA
  Arms: OA GSK4382276A Group; YA GSK4382276A Dose level 1 Group
Biological: GSK4382276A Dose level 2 — Dose level 2 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A Dose level 2 and OA GSK4382276A Selected Dose level from YA groups, at Day 1. Potential intermediate dose levels may be evaluated, with the total number of dose levels per age group not exceeding 5.
  Arms: OA GSK4382276A Group; YA GSK4382276A Dose level 2 Group
Biological: GSK4382276A Dose level 3 — Dose level 3 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A Dose level 3 and OA GSK4382276A Selected Dose level from YA groups, at Day 1. Potential intermediate dose levels may be evaluated, with the total number of dose levels per age group not exceeding 5.
  Arms: OA GSK4382276A Group; YA GSK4382276A Dose level 3 Group
Biological: GSK4382276A Dose level 4 — Dose level 4 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 4 and OA GSK4382276A Dose level 4 groups, at Day 1. Potential intermediate dose levels may be evaluated, with the total number of dose levels per age group not exceeding 5.
  Arms: YA GSK4382276A Dose level 4 Group
Biological: GSK4382276A Dose level 6 — Dose level 6 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 6 group, at Day 1.
  Arms: YA GSK4382276A Dose level 6 Group
Biological: GSK4382276A Dose level 7 — Dose level 7 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 7 group, at Day 1.
  Arms: YA GSK4382276A Dose level 7 Group
Biological: GSK4382276A Dose level 8 — Dose level 8 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 8 group, at Day 1. Potential intermediate dose levels may be evaluated with the total number of dose levels not exceeding 10 in YA and 1 in OA.
  Arms: YA GSK4382276A Dose level 8 Group
Biological: GSK4382276A Dose level 9 — Dose level 9 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 9 group, at Day 1. Potential intermediate dose levels may be evaluated with the total number of dose levels not exceeding 10 in YA and 1 in OA.
  Arms: YA GSK4382276A Dose level 9 Group
Biological: GSK4382276A Dose level 10 — Dose level 10 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 10 group, at Day 1.
  Arms: YA GSK4382276A Dose level 10 Group
Biological: GSK4382276A Dose level 11 — Dose level 11 of GSK4382276A is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA GSK4382276A level 11 group, at Day 1.
  Arms: YA GSK4382276A Dose level 11 Group
Combination Product: FDQ21A-NH — Single dose of FDQ21A-NH is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA Control 1 and OA Control groups, at Day 1.
  Arms: OA Control Group; YA Control 1 Group
Combination Product: FDQ22A-NH — Single dose of FDQ21A-NH is administered intramuscularly in the upper deltoid region of the non-dominant arm to participants in YA Control 2, at Day 1.
  Arms: YA Control 2 Group

SUMMARY:
The purpose of this first-time-in-human (FTiH) study is to assess the safety, reactogenicity and immunogenicity of GlaxoSmithKline's (GSK) messenger RNA (mRNA)-based monovalent vaccine (GSK4382276A) candidate against influenza in healthy younger adults (YA) and older adults (OA).

ELIGIBILITY:
Inclusion Criteria:

* A male or female between and including 18 and 45 years of age (YAs) or between and including 60 and 80 years of age (OAs) at the time of the study intervention administration. The age of sentinel participants in OA category will be limited to maximum 70 years.
* Healthy or medically stable participants as established by medical history, safety laboratory assessments and clinical examination.
* Body mass index ≥ 18 kg/m^2 and ≤ 32 kg/m^2.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the participant prior to performing any study-specific procedure.
* Female participants of non-childbearing potential may be enrolled in the study.
* Female participants of childbearing potential may be enrolled in the study if the participant:

  * has practiced adequate contraception for 28 days prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception for at least 1 month after study intervention administration.

Exclusion Criteria:

Medical conditions

* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or review of the participant's medical record.
* Any clinically significant* hematological coagulation or urine analysis laboratory abnormality.

  * The investigator should use his/her clinical judgement to decide which abnormalities are clinically significant.
* Current or past malignancy, unless completely resolved without sequelae for >5 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV infection, based on medical history and physical examination (no laboratory testing required).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention (including latex, poly-ethylene-glycol, egg protein and aminoglycoside antibiotics).
* Recurrent history or uncontrolled neurological disorders or seizures, including Guillain-Barré syndrome and Bell's palsy, with the exception of febrile seizures during childhood.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Significant exposure to persons with influenza or laboratory-confirmed SARS-CoV-2 within 7 days prior to Visit 1 (Day 1) and for whom a SARS-CoV-2 PCR test has not (yet) been confirmed as negative.

Prior/Concomitant therapy

* Administration of seasonal influenza vaccine within 180 days before enrollment or planned administration up to Visit 4 (Day 29).
* Administration of a vaccine not foreseen by the study protocol in the period starting 28 days before the study intervention administration, or planned administration within 28 days after the study intervention administration*, with the exception of vaccines authorized or approved for the prevention of COVID-19 (regardless of the type of vaccine).

  *In case emergency mass vaccination for an unforeseen public health threat is organized by public health authorities outside the routine immunization program, the time period described above can be reduced to 7 days, if necessary, for that mass vaccination vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified accordingly.
* Use of any investigational or non-registered product (drug, vaccine or invasive medical device) other than the study intervention during the period beginning 30 days before the study intervention administration, or their planned use during the study period.
* Administration of long-acting immune-modifying drugs within 90 days before enrollment or planned use at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the study intervention administration, or planned administration during the study period. Administration of monoclonal antibodies specifically directed against the spike protein of SARS-CoV-2 virus, for treatment of COVID-19 disease is allowed.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the study intervention administration. For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day. Inhaled, topical and intraarticular steroids are allowed.
* Previous enrolment in this study.

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions within the 1-month post-dosing period.
* History of abusive alcohol and/or drug consumption in the past 5 years.
* Any study personnel or their immediate dependents, family, or household members.
* Participants with extensive tattoos covering deltoid region on both arms that would preclude the assessment of local reactogenicity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting each solicited administration site event | From Day 1 to Day 7
  The following administration site events will be solicited: pain, redness, swelling, lymphadenopathy (defined as localized axillary, cervical or supraclavicular swelling or tenderness ipsilateral to the injection arm).
Number of participants reporting each solicited systemic event | From Day 1 to Day 7
  The following systemic events will be solicited: fever, headache, myalgia, arthralgia, fatigue, chills. Fever is defined as temperature ≥38°C/100.4°F regardless the location of measurement. The preferred location for measuring temperature is axillary.
Number of participants reporting unsolicited adverse events (AEs) | From Day 1 to Day 28
  An unsolicited AE is defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms will be reported as an unsolicited adverse event.
Number of participants reporting serious adverse events (SAEs) | From Day 1 to Day 183
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or is an abnormal pregnancy outcome.
Number of participants reporting adverse events of special interest (AESIs) | From Day 1 to Day 183
  The following events are considered as AESI in this study: severe hypersensitivity reactions within 24 hours after study intervention administration, myocarditis/pericarditis and potential immune-mediated diseases (pIMDs).
Number of participants reporting a shift from non-clinically significant laboratory value on Day 1 to clinically significant abnormal laboratory value on Day 8 or on Day 29 for hematology, clinical chemistry, coagulation and urine analysis | From Day 1 (pre-dose) to Day 8 (post-dose) or to Day 29 (post-dose)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participants condition.
Geometric mean titers (GMT) of anti-vaccine antibody titers | At Day 1
GMT of anti-vaccine antibody titers | At Day 22
Geometric mean increase (GMI) of anti-vaccine antibody titers | From Day 1 to Day 22
  GMI is defined as the geometric mean of the ratios of the post-dose anti-vaccine antibody titer over the Day 1 anti-vaccine antibody titer.
Anti-vaccine antibody titers seroconversion rate (SCR) | From Day 1 to Day 22
  SCR is defined as the percentage of dosed participants who have either an anti-vaccine antibody pre-dose titer < 1:10 and a post-dose anti-vaccine antibody titer ≥ 1:40 or a pre-dose anti-vaccine antibody titer ≥ 1:10 and at least a 4-fold increase in post-dose anti-vaccine antibody titer.
Anti-vaccine antibody seroprotection rate (SPR) | At Day 22
  SPR is defined as the percentage of dosed participants with an anti-vaccine antibody titer ≥ 1:40.

SECONDARY OUTCOMES:
GMT of anti-vaccine antibody titer. | At Day 62 and Day 183
GMI of anti-vaccine antibody titer | From Day 1 to Day 62
  GMI is defined as the geometric mean of the ratios of the post-dose anti-vaccine antibody titer over the Day 1 anti-vaccine antibody titer.
GMI of anti-vaccine antibody titer | From Day 1 to Day 183
  GMI is defined as the geometric mean of the ratios of the post-dose anti-vaccine antibody titer over the Day 1 anti-vaccine antibody titer.
Anti-vaccine antibody titer SPR | At Day 62 and Day 183
  SPR is defined as the percentage of dosed participants with an anti-vaccine antibody titer ≥ 1:40.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Belgium (2):
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
- Canada (2):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.